CLINICAL TRIAL: NCT04470336
Title: A Double-blind, Placebo-controlled, Randomized, Parallel Study to Assess the Efficacy of Collagen Supplement in Osteoarthritis
Brief Title: To Assess the Efficacy of Collagen Supplement in Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: JHB/190702/NATIVECTII/OA
Record Dates: First submitted 2020-07-08; First posted 2020-07-14 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-03

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Collagen Supplement (Active Comparator): Three capsules post-breakfast Three capsules post-dinner
  Interventions: Other: Collagen Supplement
- Glucosamine chondroitin (Other): Three capsules post-breakfast Three capsules post-dinner
  Interventions: Other: Glucosamine chondroitin
- Placebo (Placebo Comparator): Three capsules post-breakfast Three capsules post-dinner
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Collagen Supplement — Three capsules post-breakfast Three capsules post-dinner
  Arms: Collagen Supplement
Other: Glucosamine chondroitin — Three capsules post-breakfast Three capsules post-dinner
  Arms: Glucosamine chondroitin
Other: Placebo — Three capsules post-breakfast Three capsules post-dinner
  Arms: Placebo

SUMMARY:
Collagen Supplement is a natural ingredient that contains undenatured collagen derived from chicken sternum. Collagen Supplement is efficacious and safe as compared to placebo and efficacy is also comparable to glucosamine plus chondroitin for treatment of of knee Osteoarthritis

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a chronic progressive degenerative disease involving thinning of cartilage in movable joints that leads to friction between bones creating pain, stiffness, and abnormal movement. It is estimated to affect more than 20% of the population over the age of 60 years and is considered to be a major cause of morbidity, disability, and limitations on the quality of life. In India, studies have reported the prevalence of 22% to 39%, with OA being 2nd most common rheumatological disorder. , As global life expectancy increases, the prevalence of OA is expected to rise further ultimately resulting in a greater burden for healthcare. Currently, the management has largely been palliative, focusing on the alleviation of symptoms.

The principles of OA treatments primarily are to alleviate pain and stiffness and maintain function. The current treatment guidelines recommend a combination of physical therapy, use of analgesia with Acetaminophen or NSAIDs, and surgical intervention when deemed necessary. While medications slow the progression of OA and other inflammatory conditions, no proven disease-modifying agents for the treatment of knee OA currently exists. The majority of individuals are successfully managed with a combination of the aforementioned treatments, but there is still a significant group of patients in whom these treatments do not provide adequate relief. Furthermore, there remains a lack of treatments that have demonstrated effectiveness in stopping or reversing the degenerative process. , Besides, there are considerable side effects associated with the use of these drugs. As a result, OA sufferers have turned to natural nutraceuticals to ease their pain and discomfort.

In recent years, several novel agents have emerged as potential treatment alternatives to improve pain, stiffness, and function with the possibility of altering disease progression. These products are commonly used because they are well tolerated and considered safe. Among the OA patients, glucosamine and chondroitin are most commonly used and have shown to considerably reduce the pain associated with arthritis. From the nutraceutical point of view, there is a growing interest in Collagen Supplement as a solution for the treatment of OA. The Collagen Supplement has been studied extensively in both animals as well as human clinical studies. , Among animal studies, a study in the rat model of OA reported several benefits after treatment, suggesting its potential for the prevention of worsening of articular cartilage damage. In another study, porcine Collagen Supplement administration demonstrated a significant reduction of pain intensity. Also, a lower dose regimen showed meaningful pain reduction indicating its protective effect on the cartilage. Furthermore, several studies have evaluated the efficacy and safety of Collagen Supplement in individuals suffering from chronic OA. Crowley and colleagues showed that supplementation of Collagen Supplement for three months is more efficacious as compared to the combination of glucosamine plus chondroitin. In another study, 6-month administration of the Collagen Supplement significantly reduced pain, stiffness, and physical functioning as compared to glucosamine hydrochloride plus chondroitin sulfate group of participants with knee OA.

Based on the available evidence it is clear that Collagen Supplement is effective in improving joint discomfort associated with OA. Moreover, collagen products are also recognized as safe components of pharmaceutical and foods by the US Food and Drugs Administration Center for Food Safety and Nutrition. Hence, considering its symptomatic benefits, the structural effect on the cartilage and its important role in bone structure, Collagen Supplement is thought to be a viable alternative for OA patients. , Therefore, the present study aimed to evaluate the safety and efficacy of an collagen supplementation in participants suffering from knee OA. Study volunteers will be supplemented with Collagen Supplement, an collagen product for 12 weeks and assessed as per study designated efficacy and safety variables. Also, the efficacy and efficacy of Collagen Supplement will be compared with Glucosamine HCL plus chondroitin sulfate and placebo as per the set study intervals.

ELIGIBILITY:
Inclusion Criteria:

* Male & female aged ≥ 40 to ≤ 65 years suffering from knee joint pain for at least 3 months prior to screening.
* BMI ≥ 18.5 and ≤ 29.9 kg/m2.
* Non-vegetarians (Regardless of whether they eat chicken, fish, goat mutton, pork, beef or eggs).
* Screening Visual Analogue (VAS) scores for knee joint pain ≥ 60 on a 100-point scale.
* Radiographic evidence of grade II/III knee OA based on one of following criteria.
* Participants willing to stop the restricted supplements and medications prior to inclusion and throughout the study period.
* Participants willing to stop any home-based remedies or any other form of topical products intended for knee joint pain relief or any other reason for the entire study duration.
* Willing to stop the use of study designated rescue medication 48 hours prior to all assessment visits.
* Willing to abstain from food containing type II collagen only from cartilage, e.g. chicken, fish, beef, pork, etc. 48 hours prior to all assessment visits.

Exclusion Criteria:

* Prior or ongoing medical conditions (e.g. concomitant illness, psychiatric disorders, etc.), abnormal medical history or physical findings.
* Participants with history of type II diabetes and uncontrolled hypertension.
* Fasting Blood glucose > 125 mg/dl
* Systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg.
* Radiographic evidence of Grade I or Grade IV OA based on the KL radiographic criteria for osteoarthritis.
* Any history of trauma, fractures or surgery to the index joint.
* Any planned surgery (diagnostic or therapeutic intervention) to the index joint during the participation in the study.
* Participants with deformity of the knee joint.
* Participants with a diagnosed condition which may involve or involves the index joint that includes but is not limited to known rheumatic or inflammatory conditions such as rheumatoid arthritis, osteomyelitis, osteoporosis, gout, and bone metastasis.
* Other pathologic lesions on X-rays of the knee.
* Current smokers or chronic alcoholics

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-07-09 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-04-12 (Actual)

PRIMARY OUTCOMES:
modified Western Ontario and McMaster Score | Day0 Day 28 Day 56 Day 84
  Effect of consumption of IP on Joint health as assessed by the change in the (mWOMAC) total score from baseline and when compared with the placebo. [From baseline to 84 days] High score defines worst outcome and low score defines better oucome.

SECONDARY OUTCOMES:
EQ-5D-5L | Day 0 and Day 84
  Effect of consumption of IP on Joint health as assessed by the change in the EQ-5D-5L from baseline and when compared with the placebo. [From baseline to 84 days]
interleukin-6 (IL - 6) | Day 0 Day 84
  Effect of consumption of IP on Joint inflammation as assessed by the change in the inflammatory biomarker interleukin-6 (IL-6) concentration from baseline and when compared with the placebo. [From baseline to 84 days]

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shalini Srivastava, MD - Med., Study Director — Vedic Life Sciences Pvt. Ltd.
Locations (5):
- India (5):
  - Dr. Randive's knee and spine clinic, Mumbai, Maharashtra
  - PKC Hospital, Mumbai, Maharashtra
  - Dr Sonawane orthopedic clinic, Mumbai, Maharashtra
  - Rainbow Multispeciality hospital and trauma center, Navi Mumbai, Maharashtra
  - Shubham Sudbhawana Super Specialty Hospital, Varanasi, Uttar Pradesh

REFERENCES:
- [Derived] Luo C, Su W, Song Y, Srivastava S. Efficacy and safety of native type II collagen in modulating knee osteoarthritis symptoms: a randomised, double-blind, placebo-controlled trial. J Exp Orthop. 2022 Dec 23;9(1):123. doi: 10.1186/s40634-022-00559-8. PMID 36562843